CLINICAL TRIAL: NCT02218567
Title: Behavioural Problems in Huntington Disease : Analysis and Enhancement of Caregiver and Patient Experience
Acronym: HUNTEXPERT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficult
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A00327-40
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2014-06

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Interview, Psychological; Psychological Tests; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Other)
  Interventions: Behavioral: psychological interview; Behavioral: psychological tests; Other: Motor evaluation; Behavioral: Behavioral evaluation; Behavioral: cognitive tests
- Caregivers (Other)
  Interventions: Behavioral: questionnaire qualilty of life; Behavioral: psychological interview

INTERVENTIONS:
Behavioral: questionnaire qualilty of life
  Arms: Caregivers
Behavioral: psychological interview
Behavioral: psychological tests
  Arms: Patients
Other: Motor evaluation
  Arms: Patients
Behavioral: Behavioral evaluation
  Arms: Patients
Behavioral: cognitive tests
  Arms: Patients

SUMMARY:
The study hypothesis is that caregivers experience allows them to develop a lot of knowledge and know-how about behavioural problems in Huntington Disease and its consequences. The purpose of this study is to collect, describe and analyse caregivers experience in order to find and enhance their knowledge related to the adaptation to behavioural problems of Huntington Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* For patients:

  * Patients with Huntington Disease declared
  * Huntington Disease diagnosed with abnormal number of CAG repeats: 38 < nucleotide expansion (CAG)
  * Total Functional Capacity ≥ 7
  * Patients living with a caregiver
  * Aged 18 years and above
  * Subject gave its written consent
* For caregivers :

  * No risk of caregiver having Huntington disease
  * Aged 18 years and above
  * Subject gave its written consent

Exclusion Criteria:

* For patients:

  * Patient who do not live with a caregiver
  * No national health insurance affiliation
  * Being under guardianship
* For caregivers :

  * Caregiver at risk for Huntington Disease
  * No national health insurance affiliation
  * Being under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The Huntington's Disease health-related Quality of Life questionnaire | Baseline
  The primary outcome is to find a list of caregiver competences necessary to prevent and adapt to behavioural problems of Huntington Disease patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Angers, Angers, Maine Et Loire, France